CLINICAL TRIAL: NCT06715397
Title: Cross-Cultural Adaptation, Validity and Reliability of the Turkish Version of the Adolfsson-Björnsson Upper Extremity Activity Scale (ABAS) in Individuals With Upper Extremity Injuries
Brief Title: Cross-Cultural Adaptation, Validity and Reliability of the Turkish Version of the Adolfsson-Björnsson Upper Extremity Activity Scale (ABAS)
Status: Enrolling by invitation | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Dilek Hande Esen, PhD, PT, Principal Investigator, Mustafa Kemal University
Other Study IDs: E-77082166-604.01.02-809466
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Upper Extremity Injuries; Questionnaire and Survey; Reliability and Validity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with upper limb injuries: Patients with upper extremity injury, who can read and write Turkish and are between the ages of 18-64, and only participants with unchanged health status for retesting will be included in the study.
  Patients with mental and neurological disorders (major depression, schizophrenia, psychosis, stroke, cerebral palsy, etc.) and/or rheumatological disease, active local or systemic infection, cancer history, severe visual impairment, need for emergency surgery, injection in the last 3 years, sensory problems that may affect the application of scales and cognitive impairment will be excluded from the study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Activity limitation is a common problem in individuals with upper extremity disorders. Many conditions involving the shoulder complex such as traumatic and non-traumatic upper extremity pain, subacromial impingement, postoperative pain, rotator sheath tears, rotator sheath tendinopathy, shoulder arthritis, adhesive capsulitis, shoulder instabilities may lead to limitations in activities of daily living due to pain and/or symptoms. Therefore, evaluation of upper extremity activities and determination of possible limitations have an important place in the management of the disease process.

Until now, symptom-related activities of daily living in patients with upper limb disorders have often been assessed with the Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) and the Shoulder Pain and Disability Index (SPADI). However, in the development of these scales, only statements describing specific activities were used and items were not scored from easy to difficult according to activity level. There is no scale specifically developed for upper extremity pathologies that grades upper extremity activity level according to a certain level of difficulty. In order to fill this gap in the literature, Adolfsson et al. developed 'The Adolfsson-Björnsson Upper Extremity Activity Scale (ABAS)' to evaluate activities of daily living according to the perceived difficulty level in individuals with upper extremity injuries. Cross-cultural adaptation, validity and reliability of the Turkish version of the ABAS have not been studied.

The aim of this study was to make a cross-cultural Turkish adaptation of the 'The Adolfsson-Björnsson Upper Extremity Activity Scale (ABAS)' and to investigate the validity, reliability and psychometric properties of the Turkish version on individuals with upper extremity disorders.

DETAILED DESCRIPTION:
The research will be conducted at Gazi University Department of Physical Therapy and Rehabilitation, Athlete Health Unit. The research will be conducted according to the Consensus-Based Standards for the Selection of Health Measurement Instruments (COSMIN) guidelines.

Translation and cross-cultural adaptation of the ABAS will be carried out in five stages according to standard guidelines for scale translation and cross-cultural adaptation. It was planned to include 150 individuals with upper extremity disorders between the ages of 18 to 64 in the study.

The data collection for this planned study will be solely through surveys. The design of the study is a cross-sectional study aimed at developing and assessing the validity and reliability." Surveys specific to the research will be implemented in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper extremity injury, who can read and write Turkish and are between the ages of 18-64

Exclusion Criteria:

* Mental and neurological disorders (major depression, schizophrenia, psychosis, stroke, cerebral palsy, etc.) and/or rheumatological disease, active local or systemic infection, cancer history, severe visual impairment, need for emergency surgery, injection in the last 3 years, sensory problems that may affect the application of scales and cognitive impairment

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Patients with upper extremity injury, who can read and write Turkish and are between the ages of 18-64, and only participants with unchanged health status for retesting will be included in the study. Patients with mental and neurological disorders (major depression, schizophrenia, psychosis, stroke, cerebral palsy, etc.) and/or rheumatological disease, active local or systemic infection, cancer history, severe visual impairment, need for emergency surgery, injection in the last 3 years, sensory problems that may affect the application of scales and cognitive impairment will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Investigating Cross-Cultural Adaptation, Validity and Reliability of the Turkish Version of The Adolfsson-Björnsson Activity Scale (ABAS) with upper ekstremity injuries | 1 weeks
  The scale items consist of 8 different categories. The increase in the mean of the questionnaire from category 1 to 8 indicates that the upper extremity is used in higher level activities.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Hande Esen, PhD, Principal Investigator — Toros University
Locations (1):
- Toros Üniversitesi, Yenişehir, Mersi̇n, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hazar Kanik Z, Pala OO, Karabicak GO, Citaker S. Cross-cultural adaptation, validity, and reliability of the Turkish version of the Patient-Rated Elbow Evaluation. Clin Rheumatol. 2019 Nov;38(11):3289-3295. doi: 10.1007/s10067-019-04665-4. Epub 2019 Jul 6. PMID 31280380
- [Result] Langley GB, Sheppeard H. The visual analogue scale: its use in pain measurement. Rheumatol Int. 1985;5(4):145-8. doi: 10.1007/BF00541514. PMID 4048757
- [Result] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735